CLINICAL TRIAL: NCT05936242
Title: Evaluation of the INteraction Between Diet, microbiomE and Epigenetic Towards Personalized Interventions in Type 1 Diabetes (IN-DEEP Study)
Brief Title: Evaluation of Main Determinants of Postprandial Glucose Response in Type 1 Diabetes
Acronym: IN-DEEP
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, Professor, Medical Doctor, Federico II University
Other Study IDs: Prot. 338/20
Record Dates: First submitted 2023-06-30; First posted 2023-07-07 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Gut Microbiota; Dietary Habits; Postprandial Glucose Response; Hybrid artificial pancreas; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, buffy coat, feces, serum, and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to explore inter- and intra-individual determinants of postprandial glucose response in patients with type 1 diabetes using continous glucose monitoring (CGM).

Blood samples and anthropometrics will be collected during hospital visit. Participants will be asked to:

* record a seven-day food diary
* complete EPIC food frequency questionnaire
* complete questionnaires on sleep hygiene
* collect a stool sample

DETAILED DESCRIPTION:
Postprandial glucose response (PGR) is a main determinant of blood glucose control in people with type 1 diabetes (T1D) and it's still difficult to manage also in patients treated with advanced technologies. Dietary composition of meals represents one of main determinant of PGR. However, growing evidence indicates that PGR to the ingestion of the same meal may significantly differ between individuals. This effect could be explained by non-nutritional determinants, including gut microbiota composition. On this background, the aim of the study is to investigate the relative contribution of intra- and inter-individual variability in determining PGR in individuals with type 1 diabetes.

Patients with T1D regularly attending the diabetes outpatient clinic of Federico II University Teaching Hospital, will be recruited. Participants' eating habits will be collected through a 7-day food record and the European Prospective Investigation into Cancer and Nutrition (EPIC) questionnaire. Fasting blood samples will be collected for the evaluation of serum short-chain fatty acids, zonulin, metabolomic, and epigenetics. Moreover, participants will be asked to collect at home a faecal sample to determine gut microbiota composition (16s RNA sequencing). Patients will be asked to complete web-based questionnaires on sleep hygiene (Pittsburgh Sleep Quality Index, Epworth).

Postprandial glucose response will be assessed by data derived from continuous glucose monitoring (CGM) used for clinical care.

The association between the PGR, calculated as incremental AUC using the trapezoidal method, and gut microbiota composition will be assessed. Moreover, the association between PGR, dietary composition, metabolomics and epigenetics will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes

Exclusion Criteria:

* Pregnancy and/or breastfeeding
* Other chronic or acute diseases
* Use of antibiotics in the past 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals with type 1 diabetes using continuous glucose monitoring (CGM) and regularly attending the Diabetes Outpatient Clinic of Federico II University Teaching Hospital (Naples, Italy).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Postprandial glucose response | Related to 7-days food record
  Postprandial glucose response wil be calculated by the trapezoidal method as the area under the curve above the baseline value (iAUC).
  The association between iAUC and gut microbiota composition derived from the analysis of faeces samples will be assessed. The association between iAUC and energy intake and dietary composition derived from the analysis of 7-days food record and EPIC will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University Hospital, Naples, Italy

REFERENCES:
- [Derived] Abuqwider J, Pasolli E, Scida G, Corrado A, Vitale M, De Filippis F, Ercolini D, Annuzzi G, Rivellese AA, Bozzetto L. Gut microbiome profiles and associated functional pathways are linked to Mediterranean diet adherence and blood glucose control in adults with type 1 diabetes mellitus. Nutr Metab Cardiovasc Dis. 2025 Dec 2:104487. doi: 10.1016/j.numecd.2025.104487. Online ahead of print. PMID 41484024
- [Derived] Abuqwider J, Salamone D, Scida G, Corrado A, Costabile G, Luongo D, Annuzzi G, Rivellese A, Bozzetto L. Sex-specific associations of serum short-chain fatty acids with glycaemic control: an Italian cross-sectional study in adults with type 1 diabetes. BMJ Open. 2025 Mar 24;15(3):e096994. doi: 10.1136/bmjopen-2024-096994. PMID 40132856